CLINICAL TRIAL: NCT03011619
Title: Brief CBT for the Treatment of Depression During Inpatient Hospitalization
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-01404
Record Dates: First submitted 2017-01-04; First posted 2017-01-05 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Depression
Keywords: Depression; Cognitive Behavioral Therapy (CBT)
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Condition (Active Comparator): usual standard of care during an inpatient psychiatric hospitalization; medication management, group therapy, and individual therapy.
  Interventions: Behavioral: Usual Standard of Care
- CBT Condition (Experimental): If a patient is randomly assigned to the enhanced CBT group, they will participate in manualized CBT, including a sequence of sessions that builds upon prior sessions and planned exercises, including worksheets and journal entries.
  Interventions: Behavioral: Usual Standard of Care; Behavioral: Cognitive Behavioral Therapy Condition (CBT)

INTERVENTIONS:
Behavioral: Usual Standard of Care — medication management, group therapy, and individual therapy.
Behavioral: Cognitive Behavioral Therapy Condition (CBT) — CBT, including a sequence of sessions that builds upon prior sessions and planned exercises, including worksheets and journal entries.
  Arms: CBT Condition

SUMMARY:
Moderately to severely depressed subjects will be randomized to the "Control Group," who will receive care as usual, or the "CBT Group," who will receive care as usual in addition to the manualized course of Cognitive Behavioral Therapy (CBT).

DETAILED DESCRIPTION:
Participants assigned to the CBT condition will receive the usual standard of care during an inpatient psychiatric hospitalization. This includes but is not limited to medication management, group therapy, and individual therapy. If a patient is randomly assigned to the enhanced CBT group, manualized CBT, including a sequence of sessions that builds upon prior sessions and planned exercises, including worksheets and journal entries.The training M.D., who is a treating physician on HCC-10, will also intermittently and randomly observe the CBT sessions to ensure the manual properly is being followed. Although the control condition may contain elements of CBT as per the clinician completing the therapy, it is not manualized, does not include specific exercises to be completed between sessions, and is not a course that builds upon skills from the previous day, as in the CBT condition. Participants assigned to the control condition will receive the usual standard of care during an inpatient psychiatric hospitalization. This includes but is not limited to medication management, group therapy, and individual therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with depression according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria on initial assessment on the unit.
* Demonstrates at least moderate degree of depressive symptoms on MADRS, HAM-D, and CGI-S.
* Provides written informed consent.

Exclusion Criteria:

* A mental illness other than depression that is the primary cause of treatment, as determined by the Principal Investigator.
* A cognitive or neurologic disorder that inhibits ability to engage in CBT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Montgomery-Ashberg Depression Scale (MADRS) | 15 Minutes
  A ten-item clinician-administered questionnaire used to measure the severity of depressive symptoms in patients with mood disorders. The ten questions rate the severity of symptoms on scale of 0 (not present), 2 (mild), 4 (moderate), and 6 (severe). It is designed to be sensitive to change, so is often the scale of choice when interventions, such as psychotherapies, electroconvulsive therapy, or drug trials, are being studied.
Hamilton Rating Scale for Depression (HAM-D) | 20 Minutes
  Clinician-administered semi-structured interview with 17 questions. It is designed to measure the severity of depressive symptoms in patients with a primary depressive illness.
Clinical Global Impression Severity Scale (CGI-S) | 20 Minutes
  Single-item rating scale of the clinician's assessment of the global severity of depressive symptoms in relation to the clinician's total experience with depressed patients. Severity is rated on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Sergie, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- New York University School of Medicine, New York, New York, United States